CLINICAL TRIAL: NCT00201110
Title: Problem Solving & CVD Risk Management in Diabetic Blacks
Brief Title: Problem Solving and Cardiovascular Disease Risk Management in Diabetic Blacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Felicia Hill-Briggs, Principal Investigator, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 274; K01HL076644 (NIH)
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Diabetes Mellitus, Type 2; Coronary Disease
Keywords: African Americans
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Diabetes Mellitus, Type 2; Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intensive Intervention: CVD Risk Education (1 session) + Intensive Health Problem-Solving Training (8 sessions)
  Interventions: Behavioral: Problem Solving Skills
- 2 (Active Comparator): Brief Intervention: CVD Risk Education (1 session) + Brief Health Problem-Solving Training (1 session)
  Interventions: Behavioral: Problem Solving Skills

INTERVENTIONS:
Behavioral: Problem Solving Skills — Intensive Intervention: CVD Risk Self-Management Education (1 session) + Intensive Health Problem-Solving Training (8 sessions)
  Arms: 1
Behavioral: Problem Solving Skills — Brief Intervention: CVD Risk Self-Management Education (1 session) + Brief Problem-Solving Training (1 session)
  Arms: 2

SUMMARY:
The purpose of this study is to test a measurement tool and a new training intervention for problem solving in self-management of high cardiovascular disease (CVD) risk in African Americans with type 2 diabetes.

DETAILED DESCRIPTION:
BACKGROUND:

African Americans with type 2 diabetes carry a high burden of CVD risk and adverse vascular events such as stroke and peripheral vascular disease. CVD risk factors of suboptimal blood pressure, lipids, and glycemic control are controllable through medical management and lifestyle behavior modification. The traditional primary care medical management model for these chronic CVD risks is inadequate, and models are shifting toward increased disease-related decision-making and self-management on the part of the patient. Yet, precise methods for: 1) identifying patients with ineffective disease-related problem-solving skills, and 2) providing patients with disease-related education that incorporates problem-solving and decision-making skills, have yet to be determined

DESIGN NARRATIVE:

The study will test a measurement tool and a novel training intervention for problem solving as applied to self-management of high CVD risk in African Americans with type 2 diabetes. The specific aims are to: 1) assess the validity and reliability of an empirically derived assessment tool of effective versus ineffective CVD risk-related problem-solving ability (the Health Problem Solving Scale, HPSS), 2) develop a novel intervention to teach CVD risk-related problem-solving skills to ineffective problem solvers, and 3) conduct a pilot study with a sample of African Americans with type 2 diabetes who have a high CVD risk profile (suboptimal blood pressure, lipids, and/or HbA1c) AND ineffective CVD risk-related problem-solving skills, as measured by the HPSS. The principal investigator is the recipient of a Research Scientist Development Award. Her career goal is to become an independent researcher in self-management of CVD risk in high-risk African American populations, and to be a leader in the development and translation into practice of novel, theory-driven and empirically based interventions to improve patient self-management of CVD risks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes
* African American by self report
* High CVD risk profile, defined as having one or more of the following:1) suboptimal A1C (greater than 7 percent); 2) suboptimal blood pressure (SBP greater than 130 mmHg and/or DBP greater than 80 mmHg); 3) suboptimal lipid control (LDL greater than 100 mg and/or HDL less than 40 mg)
* Willing and able to give informed consent

Exclusion Criteria:

* Plan to leave area prior to study completion
* Severe diabetes complications that would interfere with the study
* End-stage disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2004-07; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
A1C | Baseline, 3-month post-intervention follow-up

SECONDARY OUTCOMES:
Barriers to Self-Management | Baseline, 1-week post-intervention follow-up, 3-month post-intervention follow-up
Dietary risk assessment | Baseline, 3-month post-intervention follow-up
Summary of Diabetes Self-Care Activities Scale | Baseline, 3-month post-intervention follow-up
Health Problem-Solving Scale | baseline, 1-week post-intervention follow-up, 3-month post-intervention follow-up
Diabetes and CVD Knowledge Test | Baseline, 1-week post-intervention follow-up, 3-month post-intervention follow-up
Blood pressure | Baseline, 3-month post-intervention follow-up
Lipid panel | Baseline, 3-month post-intervention follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Hill-Briggs, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine/General Clinical Research Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Hill-Briggs F, Gemmell L. Problem solving in diabetes self-management and control: a systematic review of the literature. Diabetes Educ. 2007 Nov-Dec;33(6):1032-50; discussion 1051-2. doi: 10.1177/0145721707308412. PMID 18057272
- [Background] Hill-Briggs F, Smith AS. Evaluation of diabetes and cardiovascular disease print patient education materials for use with low-health literate populations. Diabetes Care. 2008 Apr;31(4):667-71. doi: 10.2337/dc07-1365. Epub 2008 Jan 17. PMID 18202245
- [Background] Hill-Briggs F, Gemmell L, Kulkarni B, Klick B, Brancati FL. Associations of patient health-related problem solving with disease control, emergency department visits, and hospitalizations in HIV and diabetes clinic samples. J Gen Intern Med. 2007 May;22(5):649-54. doi: 10.1007/s11606-006-0091-2. PMID 17443373
- [Background] Hill-Briggs F, Lazo M, Renosky R, Ewing C. Usability of diabetes and cardiovascular disease education module in an African-American, diabetic sample with physical, visual, and cognitive impairment. Rehabilitation Psychology, 2008;53:1-8.
- [Background] Hill-Briggs F, Renosky R, Lazo M, Bone L, Hill M, Levine D, Brancati FL, Peyrot M. Development and pilot evaluation of literacy-adapted diabetes and CVD education in urban, diabetic African Americans. J Gen Intern Med. 2008 Sep;23(9):1491-4. doi: 10.1007/s11606-008-0679-9. Epub 2008 Jun 3. PMID 18521688
- [Result] Hill-Briggs F, Lazo M, Peyrot M, Doswell A, Chang YT, Hill MN, Levine D, Wang NY, Brancati FL. Effect of problem-solving-based diabetes self-management training on diabetes control in a low income patient sample. J Gen Intern Med. 2011 Sep;26(9):972-8. doi: 10.1007/s11606-011-1689-6. Epub 2011 Mar 29. PMID 21445680